CLINICAL TRIAL: NCT04408872
Title: A Pilot Study to Assess the Potential Value of Adding Endoscopic Ultrasound (EUS) to Esophago-gastro-duodenoscopy (EGD) in Emergency Room Patients Referred for EGD
Brief Title: EUS vs EGD in Emergency Room Patients Referred for EGD
Acronym: EUSvsEGD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not approved by the institution's scientific committee.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, A Sahai, Gastroenterologist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-9005
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Endosonography

STUDY DESIGN:
Intervention Model Description: This is an open-label two-arm, single center, superiority trial with 1:1 allocation ratio between EUS and standard intervention EGD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGD (Active Comparator): SUBJECT WILL UNDERGO ESOPHAGO-GASTRO-DUODENOSCOPY (EGD)
  Interventions: Diagnostic Test: Esophago-gastro-duodenoscopy (EGD)
- EUS (Experimental): SUBJECT WILL UNDERGO ENDOSCOPIC ULTRASOUND (EUS)
  Interventions: Diagnostic Test: Endoscopic ultrasound (EUS)

INTERVENTIONS:
Diagnostic Test: Esophago-gastro-duodenoscopy (EGD) — EGD: ENDOSCOPIC PROCEDURE DURING WHICH THE ESOPHAGUS, STOMACH AND DUODENUM ARE VISUALISED WITH A TINY CAMERA IMPLANTED AT THE END OF AN ENDOSCOPE.
  Arms: EGD
Diagnostic Test: Endoscopic ultrasound (EUS) — EUS: SAME AS EGD, BUT IN ADDITION HAS AN INTEGRATED ULTRASOUND PROBE WHICH ALLOWS TO EXAMINE THE PANCREAS, LIVER AND BILIARY SYSTEM.
  Arms: EUS

SUMMARY:
Emergency room patients referred for esophago-gastro-duodenoscopy (EGD) often have many possible causes for their symptoms. These patients inevitably undergo further testing if EGD is inconclusive, which adds costs and prolongs emergency room length of stay (LOS).EUS has traditionally been used after EGD for a myriad of reasons that no longer apply. The investigators therefore propose a prospective pilot study to determine whether adding primary EUS to EGD can reduce LOS and resource utilisation in emergency room patients referred for EGD.

DETAILED DESCRIPTION:
Emergency room patients referred for esophago-gastro-duodenoscopy (EGD) often have many possible causes for their symptoms. These inevitably undergo further testing if EGD is inconclusive, which adds costs and inevitably prolongs emergency room length of stay (LOS).

Endoscopic ultrasound (EUS) combines EGD with high-resolution ultrasound imaging of pancreas, liver and biliary system and is the best test to diagnose bile duct stones, early chronic pancreatitis, and small [<2cm] pancreatic cancers (all of which cannot be seen by regular ultrasound or CT scanning or MRI, yet are included in the differential diagnosis of EGD-negative abdominal pain).

EUS has traditionally been used after EGD, due to lack of availability, increased cost, and to increased risk due to larger scope diameter. However, the latest generation of EUS scopes have the same outer diameter as conventional gastroscopes, there is much wider availability of EUS in university and community hospital settings, and the cost per procedure is lower, due to increased procedural numbers and reduced maintenance costs.

In experienced hands, diagnostic EUS is now as safe and as accurate as EGD for diagnosing mucosal pathology and takes approximately 1 minute longer.(1; 2) Previously published work by our group suggests that EUS may reduce resource consumption in patients with unexplained abdominal pain.(3) The investigators also showed that in refractory dyspepsia with normal EGD and CT, EUS identified signs of occult chronic pancreatitis in up to 20% of cases.(4) More recently, EUS was found to identify previously undiagnosed, potential causes of unexplained abdominal pain in up to 9% of patients, or at least provides the same, if not more information than EGD and abdominal US alone.(2; 5; 6)

There are no previous studies that have prospectively compared the yield of EGD and PEUS in emergency room patients. The investigators hypothesize that adding EUS to EGD ("primary EUS" [PEUS]) can safely and more efficiently diagnose or exclude significant gastro-intestinal and pancreatico-biliary pathology in emergency room patients in whom EGD has been requested. The investigators therefore propose a prospective pilot study to perform a preliminary analysis of the potential impact of PEUS on the ability to make an early GI diagnosis (EGID), length of stay (LOS) and resource utilisation in emergency room patients referred for EGD. If there is sufficient evidence of a clinically useful impact, an appropriately powered study to determine whether PEUS is clinically superior to EGD with respect to these variables will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. EGD requested by the consulting gastroenterologist
2. Informed consent

Exclusion Criteria:

1. Evidence of hemodynamic instability and/or ongoing active GI bleeding.
2. Any suspicion of obstruction distal to the angle of Treitz.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Length of stay (LOS) at the emergency room | 48 hours
  The primary outcome will be time (hours) to discharge, or admission (for a GI diagnosis) after receipt of the endoscopy (EGD or EUS) report by the consulting gastroenterologist.

SECONDARY OUTCOMES:
Frequency of conversion to the alternate procedure (EGD to EUS, or EUS to EGD) | 48 hours
  Number of subjects who need to undergo both procedures
Alternate procedures undergone during emergency room stay | 48 hours
  Number of subsequent imaging procedures other than endoscopy
Complications during emergency room stay | 96 hours
  Defined as any event that prolongs hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: ANAND SAHAI, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (2):
- Canada (2):
  - Centre de recherche du Centre hospitalier de l'université de Montréal, Montreal, Quebec
  - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No